CLINICAL TRIAL: NCT07200544
Title: Meloxicam for Postoperative Pain in Mohs Micrographic Surgery
Brief Title: Meloxicam in Mohs Micrographic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18006
Record Dates: First submitted 2025-01-21; First posted 2025-10-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain, Acute; Skin Cancer
Keywords: Mohs micrographic surgery; Postoperative Pain; NSAID; Acetaminophen
MeSH Terms: conditions — Pain, Postoperative; Skin Neoplasms | interventions — Meloxicam; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups, and each group receives a different intervention.
Masking Description: Randomization will occur on which of the 3 groups each patient will be enrolled in, thus the investigators and participants will know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Acetaminophen/Ibuprofen) (Active Comparator): This randomized control group will take a mandatory one-time dose of 500 mg acetaminophen with alternating 200 mg ibuprofen and 500 mg acetaminophen (standard of care) every 3 hours for pain.
  Interventions: Drug: Acetaminophen 500mg
- Meloxicam 7.5 mg (Experimental): This randomly assigned experimental group will take a mandatory one-time dose of oral Meloxicam 7.5 mg with as-needed acetaminophen 500 mg every 3 hours. Administration of Meloxicam will be upon completion of Mohs closure.
  Interventions: Drug: Meloxicam 7.5 mg
- Meloxicam 15 mg (Experimental): This randomly assigned experimental group will take a mandatory one-time dose of oral Meloxicam 15 mg with as-needed acetaminophen 500 mg every 3 hours. Administration of Meloxicam will be upon completion of Mohs closure.
  Interventions: Drug: Meloxicam 15 mg

INTERVENTIONS:
Drug: Meloxicam 7.5 mg — This intervention is the mandatory oral Meloxicam 7.5mg dose after Mohs closure.
  Arms: Meloxicam 7.5 mg
Drug: Meloxicam 15 mg — This intervention is the mandatory oral Meloxicam 15mg dose after Mohs closure.
  Arms: Meloxicam 15 mg
Drug: Acetaminophen 500mg — This randomized control group will take a mandatory one-time dose of 500 mg acetaminophen with alternating 200 mg ibuprofen and 500 mg acetaminophen (standard of care) every 3 hours for pain.
  Arms: Standard of Care (Acetaminophen/Ibuprofen)

SUMMARY:
The goal of this clinical trial is to explore alternative methods of postoperative pain control in Mohs micrographic surgery. The main aims are:

* To provide more information to the Mohs surgery community regarding postoperative pain control.
* Reducing pain improves the overall comfort and well-being of patients, leading to a better post-operative experience.
* To provide patients with an alternative and potentially superior NSAID for pain control (compared to standard-of-care ibuprofen).

Researchers will compare 1) a single of dose Meloxicam 7.5 mg, followed by acetaminophen 500 mg; 2) a single dose of Meloxicam 15 mg, followed by acetaminophen 500 mg; 3) a single dose of acetaminophen 500 mg, followed by alternating ibuprofen 200 mg and acetaminophen 500 mg to see which better moderate pain control and patient satisfaction.

Participants will be asked to complete pain and patient satisfaction surveys.

DETAILED DESCRIPTION:
Mohs micrographic surgery (MMS) is a microscope-guided tissue-sparing surgical procedure for the removal of certain skin cancers, in which 100% of the surgical margin is examined. It is the gold-standard for the treatment of high-risk and aggressive nonmelanoma skin cancer. It is an incredibly safe procedure and postoperative complications are uncommon, occurring in only 0.72% of cases. It is the most cost-effective form of skin cancer removal and has higher cure rates when compared to standard excision.

Despite the safety and tolerability of the procedure, postoperative patient concerns have been assessed in the literature with pain being the most common. Using classical pain assessment models, pain is often assessed by the patient as mild to moderate. On average pain is at its worst on POD0 of surgery, with one study finding peak pain scores between 2PM to 10PM on POD02. Studies have often demonstrated that the most painful anatomical sites are the nose, ear, forehead, scalp, periorbital region, and lip with the scalp being associated with the most postoperative pain. Those who undergo linear closure or second intent healing report significantly less pain postoperatively than those who undergo flaps and full-thickness-skin grafts with age (<66 years), number of lesions, and consumption of narcotics for pain relief.

Specific Aims, long-term objectives, research accomplishments:

This study will hopefully provide more information to the Mohs surgery community regarding postoperative pain control.

Reducing pain improves the overall comfort and well-being of patients, leading to a better post-operative experience.

To provide patients with an alternative and potentially superior NSAID for pain control (compared to standard-of-care ibuprofen).

To provide a pain medication option that has a longer half-life with a reduction in patient breakthrough pain and the necessity of taking more frequent medication Discovering non-opioid pain control methods can help decrease the reliance on opioids, reducing the risk of addiction and other opioid-related side effects.

Managing pain effectively can help prevent post-operative anxiety and depression, contributing to better mental health outcomes Managing pain effectively can contribute to better Mohs surgery patient outcomes Advances in pain management can contribute to more personalized approaches, tailoring pain control strategies to individual patient needs

Background and Significance:

Standard of care postoperative pain control in Mohs micrographic surgery is alternating Tylenol and ibuprofen as directed on the manufactures label. Randomized controlled trials on postoperative pain in MMS. Upon literature review there have not been any studies in MMS using meloxicam as a postoperative pain alternative to standard of care. To date, acetaminophen and codeine, celecoxib, pregabalin, naproxen, aspirin, and other opioid prescriptions have been used for postoperative pain5-7

Meloxicam is approved for the treatment of osteoarthritis in the United States. At low doses it is COX-2 preferential, inhibiting prostanoid synthesis in inflammatory cells. In clinical trials, meloxicam was found to be as effective as naproxen, piroxicam, and diclofenac with few GI symptoms and lower incidence of perforation, obstruction and bleeding8. Compared to the medications listed above, oral meloxicam has the longest half-life at around 20 hours8. Given its long half-life, the investigators hypothesize that meloxicam will result in pain control over the postoperative time periods when pain is at its worst (POD0 and POD1). This will decrease the need for adding other pain control medicines, decrease break through pain, and increase patient satisfaction with postoperative pain control. Postoperative pain in MMS has been explored for decades and this pain-control alternative can be used as a useful tool for the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who consents to the study and are undergoing Mohs micrographic surgery at the University of Oklahoma.

Exclusion Criteria:

* Women who are pregnant, suspected to be pregnant, or planning to become pregnant during the study period will be excluded from participation.
* Chronic liver disease (chronic hepatitis, acute hepatitis, cirrhosis, NASH, NAFLD, alcoholic liver disease, hemochromatosis, Wilson's disease)
* Chronic kidney disease stage III or greater,
* Aspirin-sensitive asthma
* History of chronic NSAID use
* Patients vulnerable to drug interactions
* GI bleeds
* Peptic ulcers
* Non-English speakers

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of the use of Meloxicam vs SoC on post-operative pain levels in participants undergoing Mohs micrographic surgery. | From enrollment to suture removal, wound check or flap takedown (7-21 days)
  Pain levels at specified times post-operation (POD 0 and POD 1) will be compared among the three treatment groups. This will be collected via the Numeric Pain Scale, a 0-10 scale using descriptives faces to assess pain by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Collins, MD, Principal Investigator — University of Oklahoma, Department of Dermatology
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limthongkul B, Samie F, Humphreys TR. Assessment of postoperative pain after Mohs micrographic surgery. Dermatol Surg. 2013 Jun;39(6):857-63. doi: 10.1111/dsu.12166. Epub 2013 Mar 6. PMID 23464845
- [Background] Benzon HT. Practical management of pain. 2014;
- [Background] Evans T, Nicholas TA, Sutton AV, Wysong A. How We Do It: Postoperative Pain Control in Mohs Micrographic Surgery. Dermatol Surg. 2021 Feb 1;47(2):280-282. doi: 10.1097/DSS.0000000000002279. No abstract available. PMID 31809346
- [Background] Sniezek PJ, Brodland DG, Zitelli JA. A randomized controlled trial comparing acetaminophen, acetaminophen and ibuprofen, and acetaminophen and codeine for postoperative pain relief after Mohs surgery and cutaneous reconstruction. Dermatol Surg. 2011 Jul;37(7):1007-13. doi: 10.1111/j.1524-4725.2011.02022.x. Epub 2011 May 11. PMID 21561527
- [Background] Firoz BF, Goldberg LH, Arnon O, Mamelak AJ. An analysis of pain and analgesia after Mohs micrographic surgery. J Am Acad Dermatol. 2010 Jul;63(1):79-86. doi: 10.1016/j.jaad.2009.10.049. PMID 20542176
- [Background] Saco M, Golda N. Optimal timing of postoperative pharmacologic pain control in Mohs micrographic surgery: A prospective cohort study. J Am Acad Dermatol. 2020 Feb;82(2):495-497. doi: 10.1016/j.jaad.2019.07.077. Epub 2019 Jul 30. No abstract available. PMID 31374303
- [Background] Alam M, Ibrahim O, Nodzenski M, Strasswimmer JM, Jiang SI, Cohen JL, Albano BJ, Batra P, Behshad R, Benedetto AV, Chan CS, Chilukuri S, Crocker C, Crystal HW, Dhir A, Faulconer VA, Goldberg LH, Goodman C, Greenbaum SS, Hale EK, Hanke CW, Hruza GJ, Jacobson L, Jones J, Kimyai-Asadi A, Kouba D, Lahti J, Macias K, Miller SJ, Monk E, Nguyen TH, Oganesyan G, Pennie M, Pontius K, Posten W, Reichel JL, Rohrer TE, Rooney JA, Tran HT, Poon E, Bolotin D, Dubina M, Pace N, Kim N, Disphanurat W, Kathawalla U, Kakar R, West DP, Veledar E, Yoo S. Adverse events associated with mohs micrographic surgery: multicenter prospective cohort study of 20,821 cases at 23 centers. JAMA Dermatol. 2013 Dec;149(12):1378-85. doi: 10.1001/jamadermatol.2013.6255. PMID 24080866

DOCUMENTS (1):
  • Informed Consent Form (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT07200544/ICF_000.pdf